CLINICAL TRIAL: NCT01099046
Title: Reduction of Plasma Vasopressin Level in Patients With Meniere's Disease
Brief Title: Stress Management Therapy for Meniere's Disease
Acronym: SMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Responsible Party: Tadashi Kitahara / Associate Professor, Department of Otolaryngology & Head and Neck Surgery, Osaka University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: yk19700512
Record Dates: First submitted 2009-12-27; First posted 2010-04-06 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Meniere's Disease; Stress
Keywords: Meniere's disease; stress management; vasopressin; V2 receptor; water intake; tympanic tubing; regular sleep under dark
MeSH Terms: conditions — Meniere Disease; Diabetes Insipidus; Diabetes Insipidus, Nephrogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- medication only (No Intervention): medication = anti-diuretics
  Interventions: Behavioral: Lifestyle
- medication + water intake (Active Comparator): anti-diuretics + water intake (at least 2.0 litters per day)
  Interventions: Behavioral: Lifestyle
- medication + tympanic tubing (Active Comparator): anti-diuretics + tympanic tubing (under local anesthesia)
  Interventions: Behavioral: Lifestyle
- medication + regular sleep (Active Comparator): anti-diuretics + regular sleep (regular sleep program under dark everynight)
  Interventions: Behavioral: Lifestyle

INTERVENTIONS:
Behavioral: Lifestyle — water intake, tympanic tubing, regular sleep
  Other Names: Stress Management Therapy (SMT)

SUMMARY:
Attacks in Meniere's disease, characterized by vertigo and hearing loss, are well known to occur repeatedly under stressed environment. Hitherto, its pathology was revealed to be inner ear hydrops through human temporal bone studies in 1938. For the pathogenesis of inner ear hydrops resulting in Meniere's attacks, plasma vasopressin elevation due to stress and V2 receptor overexpression in the inner ear could be essential as a basis of this disease. In the present study, we'd like to find the effective and feasible way to reduce plasma vasopressin level in patients with Meniere's disease.

DETAILED DESCRIPTION:
BACKGROUND:

For the pathogenesis of inner ear hydrops resulting in Meniere's attacks, plasma vasopressin elevation due to stress and V2 receptor overexpression in the inner ear could be essential as a basis of this disease. In the present study, we'd like to find the effective and feasible way to reduce plasma vasopressin level in patients with Meniere's disease.

METHODS:

We estimate to enroll 200 Meniere's patients to four study groups in a randomized controlled trial at Osaka University Hospital during this study period 2010-2015. Patients are diagnosed as Meniere's patients according to the 1995 AAO-HNS criteria. Group-I consists of 50 patients who receive just traditional oral intake medication including anti-diuretics. Group-II consists of 50 patients who receive both medication and water intake (at least 2.0 litters per day). Group-III consists of 50 patients who receive both medication and tympanic tubing (under local anesthesia). Group-IV consists of 50 patients who receive both medication and sleep well (regular sleep program under dark everynight). Additional factors to medication in each group are supposed to have influence on hypothalamus. We follow up all these patients at least 12 months and evaluate stress, psychological and dizziness conditions using a couple of questionnaires. We also examine changes in plasma vasopressin level of patients in each group.

ESTIMATED RESULTS:

Through this study, we can understand the most effective and feasible way to reduce plasma vasopressin level in patients with Meniere's disease. Much more Meniere's patients may be rescued without invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as Meniere's patients according to the 1995 AAO-HNS criteria are included into this study.

Exclusion Criteria:

* Patients refused our prepared four kinds of treatments are excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Kitahara, M.D.,Ph.D., Principal Investigator — Department of Otolaryngology, Osaka University, School of Medicine
Locations (1):
- Department of Otolaryngology, Osaka University, School of Medicine, Suita, Osaka, Japan

REFERENCES:
- [Background] Kitahara T, Maekawa C, Kizawa K, Horii A, Doi K. Plasma vasopressin and V2 receptor in the endolymphatic sac in patients with delayed endolymphatic hydrops. Otol Neurotol. 2009 Sep;30(6):812-9. doi: 10.1097/MAO.0b013e3181b11db5. PMID 19638944
- [Background] Kitahara T, Doi K, Maekawa C, Kizawa K, Horii A, Kubo T, Kiyama H. Meniere's attacks occur in the inner ear with excessive vasopressin type-2 receptors. J Neuroendocrinol. 2008 Dec;20(12):1295-300. doi: 10.1111/j.1365-2826.2008.01792.x. PMID 19094077
- [Background] Kitahara T, Kubo T, Okumura S, Kitahara M. Effects of endolymphatic sac drainage with steroids for intractable Meniere's disease: a long-term follow-up and randomized controlled study. Laryngoscope. 2008 May;118(5):854-61. doi: 10.1097/MLG.0b013e3181651c4a. PMID 18520184
- [Background] Horii A, Uno A, Kitahara T, Mitani K, Masumura C, Kizawa K, Kubo T. Effects of fluvoxamine on anxiety, depression, and subjective handicaps of chronic dizziness patients with or without neuro-otologic diseases. J Vestib Res. 2007;17(1):1-8. PMID 18219099
- [Background] Horii A, Kitahara T, Uno A, Kondoh K, Morihana T, Okumura S, Nakagawa A, Mitani K, Masumura C, Kubo T. Vestibular function and vasopressin. Acta Otolaryngol Suppl. 2004 Aug;(553):50-3. doi: 10.1080/03655230410017661. PMID 15277036
- [Derived] Kitahara T, Okamoto H, Fukushima M, Sakagami M, Ito T, Yamashita A, Ota I, Yamanaka T. A Two-Year Randomized Trial of Interventions to Decrease Stress Hormone Vasopressin Production in Patients with Meniere's Disease-A Pilot Study. PLoS One. 2016 Jun 30;11(6):e0158309. doi: 10.1371/journal.pone.0158309. eCollection 2016. PMID 27362705